CLINICAL TRIAL: NCT04546438
Title: Patient Quality of Life and Safety of Treatment With Microwave Technology for Axillary Hyperhidrosis
Brief Title: Patient Satisfaction and Safety of Miradry Treatment for Axillary Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Emanuela Micu, Principal investigator, MD, PhD, Region Östergötland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FORSS-932159
Record Dates: First submitted 2020-08-29; First posted 2020-09-14 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Axillary Hyperhidrosis
Keywords: hyperhidrosis; hyperhidrosis disease severity scale (HDSS); Hospital Anxiety and Depression Scale (HADS); DLQI; HYPERHIDROSIS QUALITY OF LIFE INDEX (HidroQoL); microwave
MeSH Terms: conditions — Hyperhidrosis; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- MiraDry® treatment (Experimental): The miraDry System is a noninvasive method that utilizes microwave energy to destroy the sweat glands at the dermal-fat interface.
  Each participant will be scheduled one MiraDry ® treatment with the possiblity of a second intervention approximately three months apart if the primary objective is not fullfilled efter the first.
  Interventions: Device: miraDry®

INTERVENTIONS:
Device: miraDry® — MiraDry is a noninvasive method that uses microwave technology to destroy sweat glands.
  In this study we evaluate a higher energy level with a newer generation device, in respect with side effects and number of treatments (one or two interventions).

SUMMARY:
Primary localized hyperhidrosis is a dermatological disorder that involves excessive sweat production without an underlying cause. The disease usually affects the axillae but can also involve palms, soles of the feet or face and causes major problems in many social situations with a negative impact on quality of life and mental health.

In this study, the investigators want to investigate the effect of microwave therapy (MiraDry®) on self-rated sweating, quality of life and anxiety in participants with severe axillary hyperhidrosis. The study also aims to evaluate the safety (side effects) of the method and long term effects over 1 year of follow upp.

DETAILED DESCRIPTION:
The study is conducted during several visits or telephone follow-ups at the clinic over a period of 12 months and each patient receives a maximum of two treatments with MiraDry® (at 3-month intervals). 100 participants are planned to participate in the study.

The primary objective is to evaluate the effectiveness of the miraDry ® treatment measured by Hyperhidrosis Disease Severity Scale(HDSS).

Secondary objectives are to evaluate the side effects and the quality of Life by assessment of The Dermatology life Quality Index, The Hyperhidrosis Quality of Life Index, and Hospital Anxiety and Depression Scale.

ELIGIBILITY:
Inclusion Criteria:

* This study will recruit participants diagnosed with primarily axillary hyperhidrosis
* Informed consent is required.
* HDSS 3 or 4 (the criteria used in Sweden to allow hospital-based intervention).

Exclusion Criteria:

Participants

* who are unable to provide informed consent,
* have known allergies to lidocaine, chlorhexidine, and/or epinephrine,
* are pregnant,
* are unable to take oral antibiotics or antiseptic washes,
* have heart pacemakers or other electronic device implants,
* who need supplemental oxygen,
* have had axillary surgery procedures for hyperhidrosis,
* with previous hidradenitis suppurativa or other local infections
* had previous cancer in the treated area are not eligible to participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
The effectiveness of miraDry treatment | 1 year
  The effect of the treatment will be measured by the participants completing the Hyperhidrosis Disease Severity Scale (score 1 to 4, where a score of 3 or 4 indicates severe hyperhidrosis and a score of 1 or 2 indicates mild or moderate hyperhidrosis) att baseline (prescreening), at 3 month follow-up visit and 1 year follow-up visit.

SECONDARY OUTCOMES:
Frequency of side effects | 1 year
  Short and long term effects will be assessed during treatment and by follow -up telephone visits 2 weeks after the treatment(s), at 3 month follow-up and 1 year follow-up.
Dermatology Life Quality Index assessment | 1 year
  The participants will be asked to complete the Dermatology Life Quality Index, calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The paticipants will complete the questionnaire at baseline, at 3 months follow-up visit and 1 year follow-up visit.
Hospital anxiety and depression scale assessment | 1 year
  The participants will be asked to complete the questionnaire at baseline, at 3 months follow-up visit and 1 year follow-up visit. The questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Hyperhidrosis Quality of Life Index assessment | 1 year
  The participants will be asked to complete the Hyperhidrosis Quality of Life Index at baseline, at 3 months follow-up visit and 1 year follow-up visit. There are 18 items and score ranges from 0 to 36, with higher scores indicating a lower Hyperhidrosis Quality of Life Index.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Micu, MD PhD, Principal Investigator — Region Östergötland
Locations (1):
- Vrinnevisjukhuset, Norrköping, Sweden

IPD SHARING:
Plan to Share IPD: No